CLINICAL TRIAL: NCT05811689
Title: Trabecular Bone Score (TBS) as an Innovative Parameter Evaluation for Bone Disease's in Multiple Sclerosis (MS) Patients and Impact of Osteoporosis on the Quality of Life of Patients With MS
Brief Title: Trabecular Bone Score in Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: IRCCS Centro Neurolesi Bonino Pulejo (Other)
Responsible Party: Sponsor
Other Study IDs: TBS SM2021
Record Dates: First submitted 2023-03-17; First posted 2023-04-13 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2021-02

CONDITIONS: Multiple Sclerosis; Endocrine System Diseases; Neurologic Disorder
MeSH Terms: conditions — Multiple Sclerosis; Endocrine System Diseases; Nervous System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- sm tbs group: All patients will undergo densitometric examination with dual-energy x-ray absorptiometry (DXA) technique at our Facility.
  Interventions: Diagnostic Test: sm tbs group

INTERVENTIONS:
Diagnostic Test: sm tbs group — After collecting anthropometric data, information on environmental factors and lifestyle (smoking, alcohol intake, physical activity, sun exposure, vitamin D supplementation, fish consumption) will be acquired through a questionnaire.
  The genetic and environmental aspects related to multiple sclerosis will also be studied. Disability status will be assessed through the Kurtzke Extended Disability Status Scale (EDSS). [10] All recruited patients will be administered the questionnaire (Multiple Sclerosis Quality of Life-54 (MSQOL-54) composed of 14 scales and 54 items. The scales investigate physical functions, limitations with respect to physical and emotional role, pain, emotional well-being, degree of energy, perceptions of one's health, social, cognitive and sexual functioning, distress, changes in health, satisfaction with sexual functioning and quality of life in general.

SUMMARY:
Assess bone quality in MS patients through TBS and evaluate the potential effects exerted by different drugs used in MS treatment, which may affect BMD and TBS in MS patients

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of MS according to the latest revision of McDonald's criteria;
* patients with relapsing-remitting MS (RRMS), secondary progressive MS (SPMS) and primary progressive MS (SPMS);
* absence of cortisone therapy for at least 6 months;

Exclusion Criteria:

patients already being treated with anti-osteoporotic drugs;

• medical conditions that preclude the execution of the densitometric examination

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 300 subjects aged between 20 and 65, belonging to the MS Outpatient Clinic of the IRCCS Centro Neurolesi Bonino Pulejo will be recruited
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2021-02-14 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
DXA scanner (Horizon© DXA System) | 6 months
  The DXA scanner (Horizon© DXA System) measures bone mineral content relative to bone area.

SECONDARY OUTCOMES:
Bone Mineral Density | 6 months
  BMD will be measured in the lumbar spine (L2-L4) and in the right and left femoral neck and trochanter regions.

OTHER OUTCOMES:
TBS iNsight™ Hologic | 6 months
  A software application, the TBS iNsight™ Hologic, the analysis of the structure of the bone matrix will be carried out, in order to evaluate the quantity and quality of the microarchitecture.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Centro Neurolesi Bonino Pulejo, Messina, Italy

IPD SHARING:
Plan to Share IPD: Undecided
corresponding author